CLINICAL TRIAL: NCT01223157
Title: Saliva and Plasma Endocannabinoids Concentrations According to Feeding Status and Body Mass Index
Acronym: SALIVENDO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Jean-Pierre LEROY / Clinical Research and Innovation Director, University Hospital, Bordeaux
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CHUBX 2010/14
Record Dates: First submitted 2010-10-15; First posted 2010-10-18 (Estimated); Last update posted 2011-04-28 (Estimated); Status verified 2011-04

CONDITIONS: Obesity
Keywords: obesity; endocannabinoids
MeSH Terms: conditions — Obesity

ARMS (2):
- Obese patients (Experimental)
  Interventions: Biological: Biological data
- Normal weight subjects (Experimental)
  Interventions: Biological: Biological data

INTERVENTIONS:
Biological: Biological data — Height, Weight, waist circumference and systolic and diastolic blood pressure will be measured in obese and normal subjects. Blood and saliva sampling will be performed after an overnight fast, one hour and just before the beginning of the lunch and one hour after the end of the lunch. This will allow a measurement of fasting glycaemia and insulin, fasting cholesterol and triglycerides, liver profile. Endocannabinoids will be measured both in plasma and saliva at each time point. Gut hormones (Ghrelin and PYY) will be measured before, just before and after lunch in plasma.

SUMMARY:
Up till now, the evaluation of the endocannabinoid system (ECS) in humans needs invasive procedures. The investigators managed in the lab to determine the levels of endocannabinoids in a small number of subjects. The aim of the study is to confirm that salivary is a useful tool to evaluate the activity of the ECS both in normal weight and obese subjects that are characterised by a hyperactivity of the system. Therefore, the first objective of the study is to compare the fasting level of salivary anandamide between 12 obese patients and 12 normal weight subjects.

DETAILED DESCRIPTION:
The prevalence of obesity keeps increasing in industrialized countries. However, efficient treatments of this chronic disease are still lacking. A better understanding of the systems that regulate energy balance and eating behavior is mandatory to better understand the disease and find appropriate treatments. The endocannabinoid system (ECS) which comprises cannabinoid receptors, such as CB1 and CB2, endogenous ligands (named endocannabinoids) and specific biosynthetic and degradative pathways is a key system in the regulation of energy balance and obesity. Obesity is characterised by an hyperactivity of the system both in animal and humans. Moreover, the activity of the ECS is influenced by feeding status although only one study has only been performed in humans. The investigation of the ECS in humans needs invasive procedure (blood sampling or adipose or liver biopsy). The aim of our study is to evaluate a new tool for the ECS evaluation in humans i e the determinations of saliva concentration of endocannabinoids both in normal weight and obese subjects before and after food intake. Blood and saliva sampling will be performed after an overnight fast, one hour before, just before and one hour after a lunch in12 normal weight subjects and 12 obese characterised with anthropometric (Weight, height, BMI (Body Mass Index), waist circumference, blood pressure) and metabolic (glycaemia, insulin, lipid profile, liver profile) evaluations. The endocannabinoids concentrations will be measured with mass spectrometry in blood and saliva and gut hormones (PYY (peptide YY) and ghrelin) will be measured in plasma.

ELIGIBILITY:
Inclusion Criteria:

Obese patients :

* Age between 18 and 65 yrs
* BMI (Body Mass Index) > 30 kg/m²
* Signed inform Consent before any investigation related to the study
* No smoker

Normal weight subjects :

* Age between 18 and 65 yrs
* BMI between 18 and 25 kg/m²
* Signed inform Consent before any investigation related to the study
* No smoker

Exclusion Criteria:

* treatments that could interfere with the endocannabinoid system (anxiolytics, anticonvulsivants, antidepressants drugs)
* pregnancy, breast feeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-10; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Anandamide(AEA)concentration | Saliva sampling will be performed after an overnight fast, one hour and just before the beginning of the lunch and one hour after the end of the lunch
  The primary outcome will be the difference of fasting saliva anandamide (AEA) concentration between obese and normal weight subjects.

SECONDARY OUTCOMES:
2-AG( 2 arachidonoylglycerol), OEA (oleoylethanolamide), PEA (palmitoyléthanolamide) concentrations | Saliva sampling will be performed after an overnight fast, one hour and just before the beginning of the lunch and one hour after the end of the lunch
  to study fasting saliva concentration of 2-AG (2 arachidonoylglycerol), OEA (oleoylethanolamide), PEA(palmitoyléthanolamide) between obese and lean subjects
Food intake influence on saliva endocannabinoids | Saliva sampling will be performed after an overnight fast, one hour and just before the beginning of the lunch and one hour after the end of the lunch
  To study the effects of food intake on the levels of saliva endocannabinoids both in normal weight and obese subjects
Plasma endocannabinoids level | Blood sampling will be performed after an overnight fast, one hour and just before the beginning of the lunch and one hour after the end of the lunch
  To study the effects of food intake on the levels of plasma endocannabinoids both in normal weight and obese subjects
Correlation between saliva and plasma endocannabinoids | Blood and saliva sampling will be performed after an overnight fast, one hour and just before the beginning of the lunch and one hour after the end of the lunch
  To look for a correlation between saliva and plasma endocannabinoids
Relationship between saliva or plasma endocannabinoids and gut hormones | Blood and saliva sampling will be performed after an overnight fast, one hour and just before the beginning of the lunch and one hour after the end of the lunch
  To look for a relationship between saliva or plasma endocannabinoids and gut hormones

CONTACTS AND LOCATIONS:
Overall Officials: Blandine GATTA, Dr, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- Service of Endocrinology, Diabetology, metabolic diseases - Hôpital du Haut Lévêque - CHU de BORDEAUX, Bordeaux, France